CLINICAL TRIAL: NCT05917418
Title: Impact of Nutritional Support on Outcome,Cost/Effectiveness for Patient at Risk
Brief Title: Nutritional Support on Outcomes and Cost-effectiveness for Patients at Risk
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College (Other)
Responsible Party: Principal Investigator, Zhu-ming Jiang, Professor of General Surgery, Peking Union Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CMA2023CSPEN
Record Dates: First submitted 2023-06-03; First posted 2023-06-23 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition | interventions — Nutritional Support

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutritional support therapy group (Experimental): All participants in this group will receive proper nutritional support.
  Interventions: Dietary Supplement: nutritional support
- Routine hospital management group (No Intervention): All participants in this group will receive routine hospital management, without additional nutritional interventions.

INTERVENTIONS:
Dietary Supplement: nutritional support — nutritional support
  Arms: Nutritional support therapy group

SUMMARY:
The impact of nutritional support for the patients at nutritional risk on clinical outcomes and cost-effectiveness.

DETAILED DESCRIPTION:
Although it was often to hear that malnutrition ratio in Aisa hospitalized patient was 40%-70% , there was no evidence to elaborate the prevalence of nutritional risk and malnutrition on hospitalized patients of Asia. Also in USA no data for nutritional risk. In 2002, scientists group headed by Kondrup from : European Society for Parenteral and Enteral Nutrition demonstrated that randomized controlled clinical trials showed patients may get benefit from nutrition support when they with nutrition risk. Based on these evidences, a simpler method was established by European Society for Parenteral and Enteral Nutrition in year 2002 in Munich & it was demonstrated useful to evaluate the appropriate use of nutrition support at present time. This method was named as Nutrition Risk Screening (NRS).

Investigators propose to survey the prevalence of malnutrition & nutrition risk in large cities' large/middle size hospitalized patients in China, Europe and USA use NRS tool. As well, we also aim to figure out the current nutrition support status in current large/middle size hospitals through this survey.

Investigators also propose to evaluate the cost-effectiveness of parenteral nutrition, enteral nutrition and non-nutritional support, and to examine the clinical outcomes of nutritional support in certain patients at nutritional risk identified by NRS-2002.

For international cooperation, the partners are Professor Kondrup of Europe and Professor Nolan from Johns Hopkins Hospital,there are students from a cooperative project with Johns Hopkins Hospital for Doctor of Philosophy students 2005-2011.

ELIGIBILITY:
Inclusion Criteria:

* patients be in hospital overnight
* diagnoses according to the protocol of cohort study for cost effectiveness

Exclusion Criteria:

* patients admitting from emergency department
* patients who undergone operation before second morning of hospitalization
* patients who dose not give Informed Consents

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2026-12-01 (Estimated); Primary Completion 2040-01-30 (Estimated); Study Completion 2040-01-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of Infectious complication | during the hospital stay
  A infectious complication was defined as as the presence of recognized pathogens in body tissues that normally are sterile, confirmed by the results of culture and supported by clinical, radiologic or hematologic evidence of infection

SECONDARY OUTCOMES:
Total cost amount | during the hospital stay
  The total cost amount was considered to contain 3 items in our study. The first item was the cost of nutrition support, including nutrition solutions, nursing, physician, and other staff supervision of nutrition support preparation, administration, and catheter placement and maintenance. The second item was the cost of the infectious complication.The third item was 'other costs' associated with the hospital admission, calculated from the total costs from which the cost of nutrition support and infectious complications were subtracted.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Beijing Chest Hospital, Capital Medical University, Beijing, Beijing Municipality